CLINICAL TRIAL: NCT02468531
Title: Protection of Xenon Against Postoperative Oxygen Impairment in Adults Undergoing Stanford Type-A Acute Aortic Dissection Surgery
Brief Title: Xenon Against Postoperative Oxygen Impairment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Anzhen Hospital (Other)
Responsible Party: Principal Investigator, WeiPing Cheng, Chief physician, professor, Beijing Anzhen Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2014.7-2017.7
Record Dates: First submitted 2015-04-20; First posted 2015-06-11 (Estimated); Last update posted 2016-11-09 (Estimated); Status verified 2016-10

CONDITIONS: Acute Lung Injury
Keywords: Xenon; Standford A acute aortic dissection
MeSH Terms: conditions — Acute Lung Injury | interventions — Oxygen; Xenon

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Oxygen group (Other): 50% oxygen inhalation one hour before and after CPB,and Pulmonary Static Inflation with 50% oxygen during CPB.
  Interventions: Other: oxygen
- Xenon group (Experimental): 50% oxygen inhalation one hour before and after CPB,and Pulmonary Static Inflation with 50%,75% and 100% Xenon during CPB respectively.
  Interventions: Drug: Xenon

INTERVENTIONS:
Other: oxygen — 50% oxygen inhalation
  Arms: Oxygen group
Drug: Xenon — 50% Xenon inhalation
  Arms: Xenon group

SUMMARY:
Acute lung injury (ALI) is the vital complication of Stanford type A aortic dissection. It is confirmed that Xenon has the significant protective effect on important organs and has no suppression on the cardiovascular system. Furthermore, our earlier trial has already clarified that static inflation with 50% Xenon during cardiopulmonary bypass could attenuate ALI for Standford A acute aortic dissection. However the protection effect was restricted for the limited time. Aimed to enhance the protection effect of Xenon, we designed this randomized trial that anesthesia with 50% xenon one hour before and after CPB and pulmonary static Inflation with 50%,75% and 100% Xenon during CPB respectively.

ELIGIBILITY:
Inclusion Criteria

Consultant's clinical diagnosis of Stanford type A AAD using local pathways of diagnosis, which may include clinical history, chest radiography (X-rays), transthoracic ultrasound, and contrast-enhanced computed tomography (CT) or magnetic resonance imaging (MRI)

Patients aged 18 to 65 years

Eligible for AAD surgery

Exclusion Criteria

Have coronary heart disease, heart failure, severe cardiac tamponade, unstable hemodynamics, severe nervous system abnormalities, clinically apparent malperfusion[9] including lower limb, cerebral, coronary and renal malperfusion, and visceral ischemia, sever hepatic and renal abnormalities

Have undergone any of the cardiac and thoracic surgeries

Are unlikely to be able to perform the required clinical assessment tasks

Have significant cognitive impairment or language issues

Are unable to provide consent with regard to their participation in the study

Prescribed with non-steroidal anti-inflammatory drugs or corticosteroids before or after admission

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2015-01; Primary Completion 2017-07 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
oxygenation index | perioperative period

SECONDARY OUTCOMES:
alterations in cytokine and ROS in the perioperative period | perioperative period
extubation time | perioperative period
complications of vital organs | perioperative period

CONTACTS AND LOCATIONS:
Overall Officials: Weiping Weiping, Principal Investigator — Beijing Anzhen Hospital
Locations (1):
- Beijing Anzhen Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No